CLINICAL TRIAL: NCT05142228
Title: Erenumab as a Therapeutic Approach for the Management of Trigeminal Neuropathic Pain (TNP)
Brief Title: Erenumab-aooe for the Management of Trigeminal Neuropathic Pain.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Marcela Romero Reyes, Clinical Associate Professor, Director Brotman Facial Pain Clinic, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00097072
Record Dates: First submitted 2021-10-29; First posted 2021-12-02 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Trigeminal Neuropathy
Keywords: Trigeminal neuropathic pain; Trigeminal Nerve Injury; Idiopathic trigeminal neuralgia with continuous pain; Idiopathic painful trigeminal neuropathy; Trigeminal Nerve Diseases; Cranial Nerve Diseases; Calcitonin Gene-Related Peptide Receptor Antagonists; CGRP Receptor Antagonist; Erenumab; Neuralgia; Face Pain; Physiological effects of drugs; Trigeminal Nerve Trauma
MeSH Terms: conditions — Trigeminal Nerve Diseases; Trigeminal Nerve Injuries; Cranial Nerve Diseases; Neuralgia; Facial Pain | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erenumab-aooe (Active Comparator): Erenumab-aooe 140 mg/ml. Subcutaneous injection. Administered once every 4 weeks/28 days at visit 1, visit 2 and visit 3 for a total of 3 cycles.
  Other Name: Aimovig®
  Interventions: Drug: Erenumab-Aooe
- Placebo (Placebo Comparator): Placebo. Subcutaneous injection.Administered once every 4 weeks/28 days at visit 1, visit 2 andvisit 3 for a total of 3 cycles.
  Other name: Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Erenumab-Aooe — Administered once every 4weeks/28 days at visit 1, visit 2 and visit 3 for a total of 3 cycles.
  Other Names: Aimovig
  Arms: Erenumab-aooe
Other: Placebo — Administered once every 4weeks/28 days at visit 1, visit 2 and visit 3 for a total of 3 cycles.
  Arms: Placebo

SUMMARY:
This study is a single center, placebo-controlled, double blind, randomized, phase II pilot to evaluate the efficacy of erenumab-aooe in the management of trigeminal neuropathic pain comparing erenumab-aooe vs Placebo.

A total of 40 patients (20 each arm) aged 18-65 years old of either sex, and any race or ethnicity, presenting trigeminal neuropathic pain will be randomly assigned in a 1:1 parallel, double-blind clinical trial, to receive either Erenumab or placebo. Participants will attend 6 clinic visits (Visit 0-Visit 5) over a period of 21 weeks. Changes in pain intensity and other pain related outcomes of trigeminal neuropathic pain will be assessed. Blood samples will be collected, and participants will need to keep a daily symptom diary and answer some other questionnaires.

DETAILED DESCRIPTION:
TNP are a considerable burden and affects significantly the quality of life of the sufferer. There are medications for their management but while they may work for some patients, may not work for the others; in addition, side effects may be present for some patients with the need to decrease dosage to not optimal levels. Furthermore, the indications of these drugs are for other neuropathic pain disorders and currently there is no medication specifically indicated for the management of TNP based on its molecular pathophysiology.

The calcitonin gene-related peptide (CGRP) is a key neuropeptide involved in migraine pathophysiology. There is evidence showing that CGRP has a role in other disorders mediated by the trigeminal system in addition to migraine; CGRP has shown to have a role in orofacial pain such as in TMD and in trigeminal neuropathic pain. Erenumab-aooe is the first antibody therapeutic targeting the CGRP receptor with FDA approval for migraine prevention that is well tolerated and with a good safety profile. Therefore, the scientific premise for this study is that inhibiting the CGRP pathway in trigeminal neuropathic pain will decrease pain and pain related outcomes in a safe and well tolerated manner for this patient population.

Potential participants will be pre-screened at the Brotman Facial Pain clinic, at the Oral and Maxillofacial Surgery Clinic both at the University of Maryland, School of Dentistry, at the Pain Medicine Clinic at the University of Maryland, School of Medicine or by telephone; those willing to participate will be scheduled for a screening and baseline visit (Visit 0). During this visit, potential participants will be evaluated for eligibility for trigeminal neuropathic pain (subjects with diagnosis based on the International classification of headache disorders ICHD-3 and International classification of Orofacial Pains ICOP of idiopathic trigeminal neuralgia with concomitant continuous pain, painful posttraumatic trigeminal neuropathy or idiopathic painful trigeminal neuropathy) and written informed consent will be obtained. The screening and baseline procedures include medical history review, clinical examinations, tests and administration of questionnaires. Instructions will be given for the completion of a Daily Symptom Diary (DSD) and other questionnaires at home or online. Participants who show compliance with 80 % completion of the DSD and who meet the pain score (inclusion criteria) for 4 weeks/28 days during the baseline period from Visit 0, will be randomly assigned to one of two groups either the investigational drug or placebo and will be scheduled for Visit 1.

The study drug is Erenumab 140 mg, SC injection. Participants will attend 6 clinic visits (Visit 0-Visit 5). After randomization and on Visit 1, the participant will receive the drug or placebo. This same treatment will be administered once a month for 3 months (3 cycles/12weeks).

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all of the following criteria:

  1. Provide signed and dated informed consent form
  2. Is between 18 and 65 years of age (inclusive; male or female and any race or ethnicity)
  3. Trigeminal neuropathic pain symptoms for a minimum of 3 months prior to randomization visit, localized in any trigeminal distribution (intraoral or extraoral).
  4. Meets diagnostic criteria for Trigeminal neuropathic pain with diagnosis based on the International classification of headache disorders ICHD-3 and International classification of Orofacial Pains ICOP.

     * Diagnosed with idiopathic trigeminal neuralgia with concomitant continuous pain per ICDH-3.
     * Diagnosed with Painful posttraumatic trigeminal neuropathy or idiopathic painful trigeminal neuropathy per ICOP. May include:

       * Subjects with a history of persistent pain of idiopathic origin or after dental extractions, mandibular fracture, surgical procedure, implant procedure and root canal therapy.
  5. Participants must have a minimum mean of average daily pain intensity score of 4/10 in where 0= no pain and 10= maximum pain imaginable on a numerical rating scale (0-10), during the 4 weeks/28 days baseline period prior randomization.
  6. If taking a prescription medication daily for the management of pain (taken for at least 30 days before baseline), agrees to continue the daily use of the medication throughout the study at the same dosage.
  7. If taking prescription medication, opioid medication or OTC medications as needed or episodically for the management of pain agrees to discontinue its use prior to the Screening and Baseline Visit.
  8. If taking OTC pain medications daily agrees to continue its daily use at the same dosage throughout the study.

     • If a participant is taking an over-the-counter medication daily for management of other type of pain or for prophylaxis of myocardial infarction or stroke, the participant will be encouraged to continue the same usage of that medication throughout the study.
  9. If subjects diagnosed with migraine, are allowed only if episodic, with attacks of duration up to 5 days/month and only using triptans or NSAIDs as an abortive medication.
  10. Agrees to not start any new prescription medication for the management of trigeminal neuropathic pain or other type of pain throughout the study.
  11. Agrees to not modify their prescription regimen for current trigeminal neuropathic pain or other types of pain throughout the study
  12. Agrees not to receive any injection therapy for the management of neuropathic pain or migraine (e.g. nerve blocks, SPG blocks, steroid injections, Botox) during the course of the study
  13. Agrees not to use any neuromodulatory device for the management of neuropathic pain or migraine during the course of the study
  14. Agrees not to undergo any surgical procedure for the management of neuropathic pain during the course of the study
  15. Agrees to not use cognitive behavioral therapy (CBT), biofeedback or acupuncture for the management of pain during the course of the study.
  16. Females of childbearing potential agree to use one of the following methods of contraception throughout the study: licensed hormonal method, intrauterine device, female or male condoms with contraceptive foam, abstinence, bilateral tubal ligation/occlusion, or vasectomy in partner (if postmenopausal, must not have menstruated for at least 12 consecutive months)
  17. Willing and able to understand and comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

1. Participants with a history of congestive heart failure or uncontrolled diabetes.
2. Participants with serious hepatic, respiratory, hematologic or immunologic illnesses, an unstable cardiovascular disease, or any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or Erenumab or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the participant inappropriate for entry into this trial.
3. Participants with high blood pressure, uncontrolled high blood pressure, malignant disease, chronic constipation, any malabsorption disorders such as IBSc or any other severe acute or chronic medical or psychiatric condition (major depression, schizophrenia, dementia) or laboratory finding that may increase the risk associated with trial participation with Erenumab, that in the judgement of the investigators would interfere with study assessments and/or would make the participant inappropriate for entry into this trial.
4. Participants with active malignancy of any type or a history a malignancy (with exception of participants with malignancy surgically removed with no evidence of recurrence within 5 years before enrollment.
5. Participants with evidence or a history of drug or alcohol abuse within the past 12 months or has been diagnosed with a substance abuse disorder.
6. Participants with dental pain (determined pain of odontogenic/periodontal origin).
7. Participants with significant neurological disorders.
8. Patients with chronic migraine with and w/o aura following the ICHD-3 criteria treated or not treated with medication

   • Without excluding headache attributed to TMD
9. Participants currently taking or have previously taken Erenumab or other CGRP monoclonal antibody (mAmb) or currently taking a CGRP-Receptor antagonist (gepants) for migraine prevention.
10. Patients with hypersensitivity to Erenumab
11. Participants with trigeminal neuropathic pain taken medications for the management of trigeminal neuropathic pain in where daily dosage has been modified within three weeks before baseline.
12. Neuroimaging showing the presence of neurovascular compression or AV malformation.
13. Neuroimaging showing the presence of intracranial pathology (i.e. multiple sclerosis, tumor).
14. Presence of extracranial pathology in the area of pain (tumor, lesion).
15. Has been treated with another investigational drug or treatment within 30 days prior to the Screening and Baseline Visit
16. Has commenced a new daily prescription medication for the management of pain within 30 days prior to the Screening and Baseline Visit
17. Currently taking opioid medication whether episodically or daily, within 30 days prior to the Screening and Baseline Visit.
18. Patients sensitive to Latex
19. If planning to become pregnant, pregnant or breastfeeding.
20. Anything that, in the opinion of the investigator, would place the participant at increased risk or impede the participant's full compliance with or completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, School of Dentistry, Brotman Facial Pain Clinic, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mignogna MD, Fedele S. The neglected global burden of chronic oral diseases. J Dent Res. 2006 May;85(5):390-1. doi: 10.1177/154405910608500501. No abstract available. PMID 16632750
- [Background] Baad-Hansen L, Leijon G, Svensson P, List T. Comparison of clinical findings and psychosocial factors in patients with atypical odontalgia and temporomandibular disorders. J Orofac Pain. 2008 Winter;22(1):7-14. PMID 18351030
- [Background] Penarrocha MA, Penarrocha D, Bagan JV, Penarrocha M. Post-traumatic trigeminal neuropathy. A study of 63 cases. Med Oral Patol Oral Cir Bucal. 2012 Mar 1;17(2):e297-300. doi: 10.4317/medoral.17401. PMID 22143689
- [Background] Smith JG, Elias LA, Yilmaz Z, Barker S, Shah K, Shah S, Renton T. The psychosocial and affective burden of posttraumatic neuropathy following injuries to the trigeminal nerve. J Orofac Pain. 2013 Fall;27(4):293-303. doi: 10.11607/jop.1056. PMID 24171179
- [Background] Baad-Hansen L, Benoliel R. Neuropathic orofacial pain: Facts and fiction. Cephalalgia. 2017 Jun;37(7):670-679. doi: 10.1177/0333102417706310. Epub 2017 Apr 12. PMID 28403646
- [Background] Romero-Reyes M, Uyanik JM. Orofacial pain management: current perspectives. J Pain Res. 2014 Feb 21;7:99-115. doi: 10.2147/JPR.S37593. eCollection 2014. PMID 24591846
- [Background] International Classification of Orofacial Pain, 1st edition (ICOP). Cephalalgia. 2020 Feb;40(2):129-221. doi: 10.1177/0333102419893823. No abstract available. PMID 32103673
- [Background] Lewis MA, Sankar V, De Laat A, Benoliel R. Management of neuropathic orofacial pain. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Mar;103 Suppl:S32.e1-24. doi: 10.1016/j.tripleo.2006.10.014. PMID 17379152
- [Background] McQuay HJ, Tramer M, Nye BA, Carroll D, Wiffen PJ, Moore RA. A systematic review of antidepressants in neuropathic pain. Pain. 1996 Dec;68(2-3):217-27. doi: 10.1016/s0304-3959(96)03140-5. PMID 9121808
- [Background] McQuay H, Carroll D, Jadad AR, Wiffen P, Moore A. Anticonvulsant drugs for management of pain: a systematic review. BMJ. 1995 Oct 21;311(7012):1047-52. doi: 10.1136/bmj.311.7012.1047. PMID 7580659
- [Background] Dworkin RH, O'Connor AB, Audette J, Baron R, Gourlay GK, Haanpaa ML, Kent JL, Krane EJ, Lebel AA, Levy RM, Mackey SC, Mayer J, Miaskowski C, Raja SN, Rice AS, Schmader KE, Stacey B, Stanos S, Treede RD, Turk DC, Walco GA, Wells CD. Recommendations for the pharmacological management of neuropathic pain: an overview and literature update. Mayo Clin Proc. 2010 Mar;85(3 Suppl):S3-14. doi: 10.4065/mcp.2009.0649. PMID 20194146
- [Background] Zakrzewska JM. Medical management of trigeminal neuropathic pains. Expert Opin Pharmacother. 2010 Jun;11(8):1239-54. doi: 10.1517/14656561003767449. PMID 20426709
- [Background] Edvinsson L. The CGRP Pathway in Migraine as a Viable Target for Therapies. Headache. 2018 May;58 Suppl 1:33-47. doi: 10.1111/head.13305. PMID 29697153
- [Background] King CT, Gegg CV, Hu SN, Sen Lu H, Chan BM, Berry KA, Brankow DW, Boone TJ, Kezunovic N, Kelley MR, Shi L, Xu C. Discovery of the Migraine Prevention Therapeutic Aimovig (Erenumab), the First FDA-Approved Antibody against a G-Protein-Coupled Receptor. ACS Pharmacol Transl Sci. 2019 Sep 3;2(6):485-490. doi: 10.1021/acsptsci.9b00061. eCollection 2019 Dec 13. PMID 32259079
- [Background] Reuter U, Goadsby PJ, Lanteri-Minet M, Wen S, Hours-Zesiger P, Ferrari MD, Klatt J. Efficacy and tolerability of erenumab in patients with episodic migraine in whom two-to-four previous preventive treatments were unsuccessful: a randomised, double-blind, placebo-controlled, phase 3b study. Lancet. 2018 Nov 24;392(10161):2280-2287. doi: 10.1016/S0140-6736(18)32534-0. Epub 2018 Oct 22. PMID 30360965
- [Background] Ashina H, Iljazi A, Al-Khazali HM, Eigenbrodt AK, Larsen EL, Andersen AM, Hansen KJ, Brauner KB, Morch-Jessen T, Chaudhry B, Antic S, Christensen CE, Ashina M, Amin FM, Schytz HW. Efficacy, tolerability, and safety of erenumab for the preventive treatment of persistent post-traumatic headache attributed to mild traumatic brain injury: an open-label study. J Headache Pain. 2020 Jun 3;21(1):62. doi: 10.1186/s10194-020-01136-z. PMID 32493206
- [Background] Cady RJ, Glenn JR, Smith KM, Durham PL. Calcitonin gene-related peptide promotes cellular changes in trigeminal neurons and glia implicated in peripheral and central sensitization. Mol Pain. 2011 Dec 6;7:94. doi: 10.1186/1744-8069-7-94. PMID 22145886
- [Background] Romero-Reyes M, Pardi V, Akerman S. A potent and selective calcitonin gene-related peptide (CGRP) receptor antagonist, MK-8825, inhibits responses to nociceptive trigeminal activation: Role of CGRP in orofacial pain. Exp Neurol. 2015 Sep;271:95-103. doi: 10.1016/j.expneurol.2015.05.005. Epub 2015 May 14. PMID 25981890
- [Background] Akerman S, Romero-Reyes M. Preclinical studies investigating the neural mechanisms involved in the co-morbidity of migraine and temporomandibular disorders: the role of CGRP. Br J Pharmacol. 2020 Dec;177(24):5555-5568. doi: 10.1111/bph.15263. Epub 2020 Oct 21. PMID 32929719
- [Background] Sugawara S, Okada S, Katagiri A, Saito H, Suzuki T, Komiya H, Kanno K, Ohara K, Iinuma T, Toyofuku A, Iwata K. Interaction between calcitonin gene-related peptide-immunoreactive neurons and satellite cells via P2Y12 R in the trigeminal ganglion is involved in neuropathic tongue pain in rats. Eur J Oral Sci. 2017 Dec;125(6):444-452. doi: 10.1111/eos.12382. Epub 2017 Oct 11. PMID 29023985
- [Background] Michot B, Kayser V, Hamon M, Bourgoin S. CGRP receptor blockade by MK-8825 alleviates allodynia in infraorbital nerve-ligated rats. Eur J Pain. 2015 Feb;19(2):281-90. doi: 10.1002/ejp.616. Epub 2014 Nov 5. PMID 25370954
- [Background] Qin ZL, Yang LQ, Li N, Yue JN, Wu BS, Tang YZ, Guo YN, Lai GH, Ni JX. Clinical study of cerebrospinal fluid neuropeptides in patients with primary trigeminal neuralgia. Clin Neurol Neurosurg. 2016 Apr;143:111-5. doi: 10.1016/j.clineuro.2016.02.012. Epub 2016 Feb 10. PMID 26918582
- [Background] Farajzadeh A, Bathaie SZ, Arabkheradmand J, Ghodsi SM, Faghihzadeh S. Different Pain States of Trigeminal Neuralgia Make Significant Changes in the Plasma Proteome and Some Biochemical Parameters: a Preliminary Cohort Study. J Mol Neurosci. 2018 Dec;66(4):524-534. doi: 10.1007/s12031-018-1183-2. Epub 2018 Oct 17. PMID 30334198
- [Background] Zhang Y, Lian Y, Zhang H, Xie N, Chen Y. CGRP Plasma Levels Decrease in Classical Trigeminal Neuralgia Patients Treated with Botulinum Toxin Type A: A Pilot Study. Pain Med. 2020 Aug 1;21(8):1611-1615. doi: 10.1093/pm/pnaa028. PMID 32167549
- [Background] Tepper S, Ashina M, Reuter U, Brandes JL, Dolezil D, Silberstein S, Winner P, Leonardi D, Mikol D, Lenz R. Safety and efficacy of erenumab for preventive treatment of chronic migraine: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2017 Jun;16(6):425-434. doi: 10.1016/S1474-4422(17)30083-2. Epub 2017 Apr 28. PMID 28460892
- [Background] Ashina M, Tepper S, Brandes JL, Reuter U, Boudreau G, Dolezil D, Cheng S, Zhang F, Lenz R, Klatt J, Mikol DD. Efficacy and safety of erenumab (AMG334) in chronic migraine patients with prior preventive treatment failure: A subgroup analysis of a randomized, double-blind, placebo-controlled study. Cephalalgia. 2018 Sep;38(10):1611-1621. doi: 10.1177/0333102418788347. Epub 2018 Jul 8. PMID 29984601
- [Background] Lattanzi S, Brigo F, Trinka E, Vernieri F, Corradetti T, Dobran M, Silvestrini M. Erenumab for Preventive Treatment of Migraine: A Systematic Review and Meta-Analysis of Efficacy and Safety. Drugs. 2019 Mar;79(4):417-431. doi: 10.1007/s40265-019-01069-1. PMID 30793254
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Symonds T, Randall JA, Hoffman DL, Zakrzewska JM, Gehringer W, Lee JY. Measuring the impact of trigeminal neuralgia pain: the Penn Facial Pain Scale-Revised. J Pain Res. 2018 Jun 5;11:1067-1073. doi: 10.2147/JPR.S152958. eCollection 2018. PMID 29892203
- [Background] Von Korff M, Ormel J, Keefe FJ, Dworkin SF. Grading the severity of chronic pain. Pain. 1992 Aug;50(2):133-149. doi: 10.1016/0304-3959(92)90154-4. PMID 1408309
- [Background] Perrot S, Lanteri-Minet M. Patients' Global Impression of Change in the management of peripheral neuropathic pain: Clinical relevance and correlations in daily practice. Eur J Pain. 2019 Jul;23(6):1117-1128. doi: 10.1002/ejp.1378. Epub 2019 Mar 18. PMID 30793414
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Svensson P, Drangsholt M, Pfau DB, List T. Neurosensory testing of orofacial pain in the dental clinic. J Am Dent Assoc. 2012 Aug;143(8):e37-9. doi: 10.14219/jada.archive.2012.0301. No abstract available. PMID 22855909
- [Background] Kim HJ, Greenspan JD, Ohrbach R, Fillingim RB, Maixner W, Renn CL, Johantgen M, Zhu S, Dorsey SG. Racial/ethnic differences in experimental pain sensitivity and associated factors - Cardiovascular responsiveness and psychological status. PLoS One. 2019 Apr 18;14(4):e0215534. doi: 10.1371/journal.pone.0215534. eCollection 2019. PMID 30998733
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Background] Nasri-Heir C, Khan J, Benoliel R, Feng C, Yarnitsky D, Kuo F, Hirschberg C, Hartwell G, Huang CY, Heir G, Korczeniewska O, Diehl SR, Eliav E. Altered pain modulation in patients with persistent postendodontic pain. Pain. 2015 Oct;156(10):2032-2041. doi: 10.1097/j.pain.0000000000000265. PMID 26098442
- [Background] Sarnthein J, Stern J, Aufenberg C, Rousson V, Jeanmonod D. Increased EEG power and slowed dominant frequency in patients with neurogenic pain. Brain. 2006 Jan;129(Pt 1):55-64. doi: 10.1093/brain/awh631. Epub 2005 Sep 23. PMID 16183660
- [Background] de Vries M, Wilder-Smith OH, Jongsma ML, van den Broeke EN, Arns M, van Goor H, van Rijn CM. Altered resting state EEG in chronic pancreatitis patients: toward a marker for chronic pain. J Pain Res. 2013 Nov 25;6:815-24. doi: 10.2147/JPR.S50919. PMID 24379694
- [Background] Seminowicz DA, Bilska K, Chowdhury NS, Skippen P, Millard SK, Chiang AKI, Chen S, Furman AJ, Schabrun SM. A novel cortical biomarker signature for predicting pain sensitivity: protocol for the PREDICT longitudinal analytical validation study. Pain Rep. 2020 Jul 27;5(4):e833. doi: 10.1097/PR9.0000000000000833. eCollection 2020 Jul-Aug. PMID 32766469
- [Background] Furman AJ, Thapa T, Summers SJ, Cavaleri R, Fogarty JS, Steiner GZ, Schabrun SM, Seminowicz DA. Cerebral peak alpha frequency reflects average pain severity in a human model of sustained, musculoskeletal pain. J Neurophysiol. 2019 Oct 1;122(4):1784-1793. doi: 10.1152/jn.00279.2019. Epub 2019 Aug 7. PMID 31389754
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Bazanova OM, Vernon D. Interpreting EEG alpha activity. Neurosci Biobehav Rev. 2014 Jul;44:94-110. doi: 10.1016/j.neubiorev.2013.05.007. Epub 2013 May 20. PMID 23701947
- [Background] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Background] Gomez-Arguelles JM, Dorado R, Sepulveda JM, Herrera A, Arrojo FG, Aragon E, Huete CR, Terron C, Anciones B. Oxcarbazepine monotherapy in carbamazepine-unresponsive trigeminal neuralgia. J Clin Neurosci. 2008 May;15(5):516-9. doi: 10.1016/j.jocn.2007.04.010. Epub 2008 Apr 2. PMID 18378142
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Son H, Friedmann E, Thomas SA. Application of pattern mixture models to address missing data in longitudinal data analysis using SPSS. Nurs Res. 2012 May-Jun;61(3):195-203. doi: 10.1097/NNR.0b013e3182541d8c. PMID 22551994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited and pre-screened at the Brotman Facial Pain clinic, University of Maryland, School of Dentistry.
  05/31/2022 was the date of the first participant enrolled. Enrollment period: 05/31/2022 to 10/21/2022
  Total number of subjects prescreened: 9
Pre-assignment Details: 5 participants signed consent and enrolled.
  1 completed study; 1 was found ineligible short after consent/enrollment due to medical history update; 1 lost follow up after baseline visit; 1 lost follow up after enrollment; 1 was dis-enrolled due to study closure.
  Baseline period consisted of 28 days/4 weeks prior randomization. Only one participant was assigned (blind/randomized) to one arm/group.
Groups:
- Erenumab-aooe: Erenumab-aooe 140 mg/ml. Subcutaneous injection. Administered once every 4 weeks/28 days at visit 1, visit 2 and visit 3 for a total of 3 cycles.
  Other Name: Aimovig®
  Erenumab-Aooe: Administered once every 4weeks/28 days at visit 1, visit 2 and visit 3 for a total of 3 cycles.
- Placebo: Placebo. Subcutaneous injection.Administered once every 4 weeks/28 days at visit 1, visit 2 andvisit 3 for a total of 3 cycles.
  Other name: Placebo
  Placebo: Administered once every 4weeks/28 days at visit 1, visit 2 and visit 3 for a total of 3 cycles.
Period: Overall Study
Arm/Group | Erenumab-aooe | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed baseline period and randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erenumab-aooe | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change of >= 30% Reduction in the Monthly (28 Days) Average Pain Score From Baseline to Visit 4, Compared to Placebo.
Description: Assessment of the efficacy of erenumab-aooe in the proportion of participants that achieve >=30% reduction (Yes/no) in monthly (28 days) average pain score from baseline to Visit 4 (the last monthly treatment cycle), compared to placebo. The daily pain intensity score will be measured on a 11-point (0-10) numeric rating scale (NPRS) and reported in the Daily Symptom Diary (DSD). The monthly mean pain intensity score will be determined from baseline (4 weeks/28 days), for each month during the 12 weeks of treatment.
Time Frame: From Visit 0 (Baseline phase/Study day 0) to Visit 4 (Study day 112 +/- 7)
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Efficacy of Erenumab-aooe Compared to Placebo on the Reduction in Monthly Average Daily Pain Score From Baseline to the End of 12-week Treatment Period.
Description: Comparison of erenumab-aooe with placebo in the reduction of pain score from baseline continuously through to the end of 12 weeks (Visit 4).
Time Frame: From Visit 0 (Baseline phase/Study day 0) to Visit 4 (study day 112 +/- 7)
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change of >= 30% Reduction in the Monthly (28 Days) Average Pain Score Compared to Placebo From Baseline to Visit 5.
Description: Assess the efficacy of erenumab-aooe compared to placebo on the proportion of subjects who achieved a least 30% reduction in the monthly average daily pain score from baseline to Visit 5 (follow-up/final visit).
Time Frame: From Visit 0 (Baseline phase/Study day 0) to Visit 5 ( study day 140 +/- 7)
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Participant Ratings Compared to Placebo for Improving Physical Function and Health Related Quality of Life in Patients With Trigeminal Neuropathic Pain Measured by the Penn Facial Pain Scale-Revised.
Description: Efficacy of erenumab-aooe compared to placebo in improvement on burden/disability of daily activities related to trigeminal neuropathic pain (e.g. chewing, eating, talking, touching) measured by the Penn Facial Pain Scale-Revised. 12 items. The higher the score the more pain and disability.
Time Frame: Visit 0 (baseline/study day 0), Visit 1 (study day 28), Visit 2 (study day 56), Visit 3 (study day 84), Visit 4 (study day 112) and Visit 5 (140) +/- 7
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Graded Chronic Pain Scale (GCPS) Outcomes During Erenumab-aooe Treatment, After Treatment and Compared to Placebo.
Description: The GCPS includes 7 items and assesses 2 dimensions of pain, pain intensity and pain-related disability. A higher grade means a worse outcome.
Time Frame: as for outcome 4
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in the Hospital Anxiety and Depression Scale (HADS). Anxiety and Depression Score Change During Erenumab-aooe Treatment, After Treatment and Compared to Placebo.
Description: The HADS evaluates anxiety (7 items) and depression (7 items) with a 14-item instrument assessing symptoms on a 4-point scale rated from 0 "not at all" to 3 "very often indeed". Responses provide separate scores for anxiety and depression. A higher score means a worse outcome.
Time Frame: as for outcome 4
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Impression of Overall Status Measured by the Patient Global Impression of Change (PGIC) During Erenumab-aooe Treatment, After Treatment and Compared to Placebo.
Description: The PGIC measures change in participant's overall status on a scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: as for outcome 4
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Change of Pro-inflammatory and Anti-inflammatory Cytokine Profiles (Th1/Th2) When Compared to Placebo.
Description: Blood samples will be evaluated for the presence of proinflammatory and anti-inflammatory cytokines.
Time Frame: Visit 0 (Baseline/study day 0) and Visit 4 (study day 112) +/- 7
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Change in Nociceptive Processing and Sensitization Determined With Quantitative Sensory Testing (QST) Measurements When Compared to Placebo.
Description: Assessment of erenumab-aooe influence in nociceptive processing and sensitization determined with QST measurements.
Time Frame: Visit 0 (Baseline/Study day 0) and Visit 4 (study day 112 +/- 7)
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Change in Pain Sensitivity Determined by Peak Alpha Frequency (PAF) Measurements During EEG (Electroencephalogram) Assessment When Compared to Placebo.
Description: Assessment of erenumab-aooe influence in pain sensitivity determined by PAF measurements during EEG assessment.
Time Frame: Visit 0 (Baseline/Study day 0) and Visit 4 (study day 112 +/- 7)
Population: Only one subject was randomly blinded and assigned to study drug (Erenumab-aooe). Data were not collected to report.
Arm/Group | Erenumab-aooe | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 weeks
Description: No participants were recruited to the Placebo Arm
Arm/Group | Erenumab-aooe | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to low enrollment rate. Ultimately we only had one participant in only one group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT05142228/Prot_SAP_001.pdf